CLINICAL TRIAL: NCT02936245
Title: Predictors of Outcome and Natural History in Patients With Cervical Spondylotic Myelopathy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: PONH CSM
Record Dates: First submitted 2016-10-12; First posted 2016-10-18 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Cervical Spondylosis With Myelopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: no specific intervention — We will not assign specific intervention in this research. We will record their baseline characteristics, received treatment, and assess the outcomes to analysis the predictors of outcome and natural history in patients with cervical spondylotic myelopathy.

SUMMARY:
Cervical spondylotic myelopathy (CSM) is the most frequent cause of myelopathy in those over the age of 50. They claim that surgical treatment of myelopathy, especially of the mild and moderate forms, has not shown better results than conservative treatment in the long term, and criteria for the indication and the timing of the operation have not been established. In order to get some more reliable data, a long-term follow up observational study will be started to confirm the effects of long term for conservative treatment.

DETAILED DESCRIPTION:
Cervical spondylotic myelopathy (CSM) is the most frequent cause of myelopathy in those over the age of 50 [1]. It is believed to have a generally progressive course over a period of years, with sudden acceleration especially following a slight head and neck injury, leading to significant disability [2, 3]. The treatment of CSM remains a problem, particularly in the mild and moderate forms without rapid progression.

Excellent outcomes for surgery have been presented in many studies. All of the studies, however, are retrospective, and many lack a clear design, standard criteria, control groups, and sufficient follow-up, so it is difficult to compare [4, 5, 6]. Furthermore, several studies and critical reviews are not so optimistic. They claim that surgical treatment of myelopathy, especially of the mild and moderate forms, has not shown better results than conservative treatment in the long term, and criteria for the indication and the timing of the operation have not been established [7, 8, 9]. Twenty-five percent of patients with laminoplasty suffer from severe neck and shoulder pain for more than 3 months [10], with significant morbidity from the iliac crest donor site etc. Surgery to decompress and stabilize the spine is often advocated for severe or progressive symptoms, with mixed results. About two-thirds of patients improve with surgery, whereas surgery is not successful in 15% to 30% of cases [11].

In order to get some more reliable data, a long-term follow up observational study will be started to confirm the effects of long term for conservative treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical signs and symptoms of cervical cord dysfunction
2. Magnetic resonance imaging (MRI) criteria for cervical multisegmental cord compression and/or myelopathy due to spondylosis (including soft disc herniations) with or without developmentally narrow spinal canal
3. Age under 75 years
4. Patient's consent to conservative treatment It has been suggested that magnetic resonance imaging

Exclusion Criteria:

1. Spinal cord compression, without clinical symptoms
2. Previous surgery on the cervical spine
3. Uncertainty about the presence of significant additional diseases (such as Motor neurone disease, progressive polyarthritis)
4. Cervical cord dysfunction due to tumors, trauma, soft disc herniation or previous surgery
5. Serious that require a surgical procedure

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cervical spondylosis myelopathy caused by spondylosis (including soft disc herniations) with or without developmentally narrow spinal canal
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2013-10; Primary Completion 2019-12 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Japanese Orthopaedic Association scale | 3 years
  Japanese Orthopaedic Association scale assessed for 3 years

SECONDARY OUTCOMES:
Adverse Event | 6 months, 1, 2, 3,4 and 5 years
  Adverse Event recorded 6 months, 1, 2, 3,4 and 5 years
Visual Analogue Scale | 6 months, 1, 2, 3,4 and 5 years
  Visual Analogue Scale assessed for 6 months, 1, 2, 3,4 and 5 years
the Medical Outcomes Study short form health survey-36 | 6 months, 1, 2, 3,4 and 5 years
  assessed for 6 months, 1, 2, 3,4 and 5 years
Neck Disability Index | 6 months, 1, 2, 3,4 and 5 years
  Neck Disability Index assessed for 6 months, 1, 2, 3,4 and 5 years
Japanese Orthopaedic Association scale | 6 months, 1, 2, 4 and 5 years
  Japanese Orthopaedic Association scale assessed for 6 months, 1, 2, 3,4 and 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Wang Yongjun, PhD, Study Chair — Longhua Hospital, Shanghai Universiy of Traditional Chinese Medicine
Locations (1):
- Longhua Hospital, Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
individual participant data (IPD) available

REFERENCES:
- [Result] Young WF. Cervical spondylotic myelopathy: a common cause of spinal cord dysfunction in older persons. Am Fam Physician. 2000 Sep 1;62(5):1064-70, 1073. PMID 10997531
- [Result] Law MD Jr, Bernhardt M, White AA 3rd. Cervical spondylotic myelopathy: a review of surgical indications and decision making. Yale J Biol Med. 1993 May-Jun;66(3):165-77. PMID 8209553
- [Result] Rowland LP. Surgical treatment of cervical spondylotic myelopathy: time for a controlled trial. Neurology. 1992 Jan;42(1):5-13. doi: 10.1212/wnl.42.1.5. PMID 1734322
- See also: Cervical spondylotic myelopathy: a common cause of spinal cord dysfunction in older persons — https://www.ncbi.nlm.nih.gov/pubmed/10997531
- See also: Cervical spondylotic myelopathy: a review of surgical indications and decision making. — https://www.ncbi.nlm.nih.gov/pubmed/?term=Cervical+spondylotic+myelopathy%3A+a+review+of+surgical+indications+and+decisions+making
- See also: Surgical treatment of cervical spondylotic myelopathy: time for a controlled trial — https://www.ncbi.nlm.nih.gov/pubmed/1734322
- See also: Cervical spondylotic myelopathy: a review of surgical indications and decision making — https://www.ncbi.nlm.nih.gov/pubmed/?term=Cervical+spondylotic+myelopathy%3A+a+review+of+surgical+indications+and+decisions+making